CLINICAL TRIAL: NCT05705791
Title: Clinical Investigation Evaluating Safety and Efficacy of Selective Intra-arterial 166Holmium Radiation Therapy in Combination With Atezolizumab and Bevacizumab for Non Resectable Hepatocellular Carcinoma
Acronym: HOLMBRAVE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-001749-19; 2021/3330 (Other: CSET number)
Record Dates: First submitted 2023-01-17; First posted 2023-01-31 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Simon's two stage design: In the first stage, 23 evaluable patients will be accrued. If there are 7 or fewer responses (complete or partial response) in these 23 patients, the clinical investigation will be stopped for futility. Otherwise, 10 additional evaluable patients will be accrued for a total of 33.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 166Holmium SIRT arm (Experimental): 166Holmium selective internal intra-arterial radiation therapy (QuiremSpheres®, experimental medical device) in combination with approved first line therapy:
  * Atezolizumab1200mg Q3W IV
  * Bevacizumab 15mg/kg Q3W IV
  Interventions: Device: QuiremSpheres

INTERVENTIONS:
Device: QuiremSpheres — 166Holmium selective internal intra-arterial radiation therapy at C1D15 of the Atezolizumab and Bevacizumab therapy
  Other Names: 166Holmium microspheres; 166Holmium SIRT

SUMMARY:
The goal of this clinical trial is to evaluate the added value of 166Holmium SIRT to Atezolizumab-Bevacizumab in patients with non resectable HCC. The primary endpoint is the Best Objective Response Rate at 6 months after 166Holmium SIRT according to mRECIST.

Participants will be treated by :

* Approved first line systemic therapy: Atezolizumab (1200mg Q3W, IV) with Bevacizumab (15mg/kg Q3W, IV)
* In combination with 166Holmium selective internal intra-arterial radiation therapy (Quirem Spheres®, the investigational medical device) after a work-up phase considered as "favorable".

Participants will be followed up to 12 months after the first cycle of Atezolizumab and Bevacizumab therapy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years old
* Patient should understand, sign, and date the written informed consent form prior to any investigation-specific procedures performed.
* Patient should be able to comply with investigational procedure, tissue and blood sample collection and willing to comply with investigation visits and procedures as per clinical investigation plan.
* Patients must have pathological confirmation of HCC.
* HCC classed Barcelona Clinic Liver Cancer (BCLC) stage C
* Patient should be considered as non resectable by Multidisciplinary Team and liver surgeon, and non-eligible for liver transplantation
* Patient should be eligible for 1st line Atezolizumab and Bevacizumab combination therapy. Patients previously treated by a local therapy are eligible.
* Patient with active intrahepatic HCC.
* Patients with or without active viral infection (i.e., HCV, HBV) are eligible. In case of active hepatitis B, the patient should be treated with an anti-HBV therapy during the investigational procedure.
* Patients should have measurable disease as defined by mRECIST criteria for response assessment.
* ECOG status of 0 or 1 (Appendix 2).
* Life expectancy of ≥ 12 weeks at the time of informed consent per Investigator assessment.
* Adequate organ function as defined by the following:

  1. White blood cells (WBCs) ≥ 2000/mL
  2. Platelets ≥ 70 × 103/mL
  3. Hemoglobin ≥ 8.0 g/dL
  4. Creatinine < 1.5 × ULN or creatinine clearance ≥ 40mL/min (Cockcroft-Gault formula)
  5. ALT and AST ≤ 3 × ULN
  6. Lipase and amylase ≤ 1.5 × ULN
  7. Total bilirubin ≤ 1.5 × ULN
* Child-Pugh A, Without history of encephalopathy or clinically significant ascites
* Women of childbearing potential (WOCBP) must have a negative urine or serum β-HCG pregnancy test within 7 days prior registration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Sexually active female patients must agree to use two methods of effective contraception*, one of them being a barrier method, or to abstain from sexual activity during the clinical investigation and for at least 6 months after last drug administration of the investigational procedure or must refrain from heterosexual activity during this same period**.

  * Acceptable contraceptive methods include single or combined contraceptive methods that result in a failure rate of < 1% per year, such as: tubal ligation, male sterilization, hormonal implants, proper use of combined oral or injected hormonal methods (e.g., two barrier methods such as a condom and a cervical cap) may be combined to achieve a failure rate of < 1% per year. Barrier methods must always be supplemented with the use of a spermicide.

  ** Abstinence is acceptable only if it is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* Sexually active males patients must agree to use condom during the clinical investigation and for at least 7 months after the last drug administration of the investigational procedure. Also, it is recommended the childbearing potential female partner uses a highly effective method of contraception for the same duration.
* Patients shall be eligible to undergo pre-treatment and on-treatment tumor biopsies. Patients who either do not consent to a pre-treatment tumor biopsy or do not have accessible lesions will not be eligible.
* Patients must be affiliated to a social security system or beneficiary of the same

Exclusion Criteria:

* Patients with a prior malignancy are excluded, except those with prior malignancies treated more than 2 years previously (at the time of informed consent) with curative intent with no evidence of disease during the interval and who are considered by the Investigator to present a low risk for recurrence, will be eligible.
* A known or underlying medical condition that, in the opinion of the Investigator, could make the administration of investigational procedure combination hazardous to the subject or could adversely affect the ability of the subject to comply with or tolerate clinical investigation.
* Requirement for daily supplemental oxygen
* Previous external radiation therapy to the liver
* Uncorrectable abnormal vascular anatomy at pre-assessment angiogram that would result in significant reflux to of hepatic arterial blood to the lung, stomach, pancreas or bowel
* Complete main portal vein thrombosis
* History or active autoimmune disease with the following exceptions: patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone, patients with controlled Type 1 diabetes mellitus on a stable insulin regimen and patients with mild autoimmune skin disorders (such as eczema or atopic dermatitis involving <10% of the skin) may be eligible for this clinical investigation
* Any of the following within the 6 months prior to clinical investigation entry: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack.
* A confirmed history of encephalitis, meningitis, or uncontrolled seizures in the year prior to informed consent.
* Positive blood screen for human immunodeficiency virus (HIV) with acquired immunodeficiency syndrome (AIDS). Patients with controlled HIV infection under anti-retroviral therapy and normal CD4+ T-cell counts (>500/mm3) could be considered eligible by the investigator if the patient fulfills the other inclusion/exclusion criteria.
* Evidence of active infection that requires systemic antibacterial, antiviral, or antifungal therapy ≤ 7 days prior to inclusion.
* Any other significant acute or chronic medical illness. Any other sound medical, psychiatric, and/or social reason as determined by the Investigator.
* Subjects who are unable to undergo and/or tolerate venous AND arterial access (evaluated on pre-treatment imaging)
* Patients that have received within 4 weeks or 5 half-lives (whichever is shorter) from inclusion and who are planned to receive the following during investigational procedure:

  * Any other investigational drug
  * Any anticancer therapy (chemotherapy, biologics, therapeutic vaccines, radiotherapy, or hormonal treatment).
  * Treatment with capecitabine within two months prior to treatment, or patient who will be treated with capecitabine at any time following treatment with QuiremSpheres®
  * Concomitant use of herbal therapies/traditional Chinese medicine with anti-cancer activity included in the label is not permitted because of potential drug-drug interactions.
  * Vaccines containing replicating live virus
  * Allergen hyposensitization therapy
  * Growth factors, e.g., granulocyte-colony stimulating factor (G-CSF), granulocyte macrophage-colony stimulating factor (GM-CSF), erythropoietin
  * Major surgery. The patient must recover from any major surgical operations before being treated with QuiremSpheres.
  * Bisphosphonates or anti-RANKL therapy
  * Systemic corticosteroids or other systemic immunosuppressive medications. The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) is allowed.
  * Coumadin or warfarin are prohibited. The use of LMWH is allowed.
  * Local treatments on the targeted tumors (percutaneous ablations, chemoembolization, radiation therapy, or liver surgery).
* Previous allogeneic hematopoietic stem cell transplantation or previous solid organ transplantation requiring systemic immunosuppressive therapy
* History of severe allergy, anaphylactic or other hypersensitivity reactions to chimeric or humanized antibodies or to biopharmaceutical produced in Chinese hamster ovarian cells or to any components of the drugs of the investigational procedure
* Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent
* Pregnant or breastfeeding women or intending to become pregnant during the clinical investigation.
* Patients with untreated or incompletely treated varices with bleeding or high-risk for bleeding. Patients must undergo an esophagogastroduodenoscopy (EGD), and all size of varices (small to large) must be assessed and treated per local standard of care prior to enrollment. Patients who have undergone an EGD within 6 months of prior to initiation of investigational procedure (D1C1 of the Atezolizumab/Bevacizumab therapy) do not need to repeat the procedure.
* Inadequately controlled arterial hypertension (defined as systolic blood pressure (BP) > or = 150 mmHg and/or diastolic blood pressure > 100 mmHg), based on an average of > or = 3 BP readings on > or = 2 sessions
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to initiation of investigational procedure (D1C1 of the Atezolizumab/Bevacizumab therapy)
* History of hemoptysis (> or = 2.5 mL of bright red blood per episode) within 1 month prior to initiation of investigational procedure (D1C1 of the Atezolizumab/Bevacizumab therapy)
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Any other contraindication to the experimental medical device use :

  * ascites or are in clinical liver failure;
  * significantly abnormal synthetic and excretory liver function tests (LFTs);
  * a lung dose exceeding 30 Gy in a single treatment;
  * uncorrectable extrahepatic deposition. Activity in the falciform ligament, portal lymph nodes and gallbladder is accepted.
* History of hypersensitivity reactions to the active substance of 99mTc-MAA or to one of its excipients or to one of the components of the radiolabeled pharmaceutical.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | at 6 months after intervention
  complete or partial response

SECONDARY OUTCOMES:
Type of treatment related adverse events (AEs) and adverse device effects (ADEs) | from start of treatment to 100 days after the administration of SIRT
  regarding to NCI-CTCAE v5.0
Frequency of treatment related adverse events (AEs) and adverse device effects (ADEs) | from start of treatment to 100 days after the administration of SIRT
  regarding to NCI-CTCAE v5.0
Severity of treatment related adverse events (AEs) and adverse device effects (ADEs) | from start of treatment to 100 days after the administration of SIRT
  regarding to NCI-CTCAE v5.0
Progression Free Survival (PFS) | at 12 weeks, at 6 months and at 12 months
  Evolution of Progression Free Survival (PFS)
Liver PFS | at 12 weeks, at 6 months and at 12 months
  Evolution of liver PFS
Overall Survival (OS) | at 12 weeks, at 6 months and at 12 months
  Evolution of Overall Survival (OS)
Objective Response Rate (ORR) | at 12 weeks, at 6 months and at 12 months
  Evolution of Objective Response Rate (ORR)
Evaluate alternative response evaluation criteria | from start of treatment to last follow-up visit
  iRECIST, itRECIST

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - AP-HP Hôpital Beaujon, Clichy
  - Centre Georges-François Leclerc, Dijon
  - CHU François Mitterand, Dijon
  - Hôpital Saint Eloi, Montpellier
  - CHU Nantes, Nantes
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No